CLINICAL TRIAL: NCT02888236
Title: LEO 32731 for the Treatment of Moderate to Severe Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0058-1072
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 32731 tablet (Experimental): LEO 32731 30 mg two times daily for 16 weeks
  Interventions: Drug: LEO 32731
- LEO 32731 Placebo tablet (Placebo Comparator): LEO 32731 placebo two times daily for 16 weeks
  Interventions: Drug: LEO 32731 Placebo

INTERVENTIONS:
Drug: LEO 32731
  Arms: LEO 32731 tablet
Drug: LEO 32731 Placebo
  Arms: LEO 32731 Placebo tablet

SUMMARY:
A study of LEO 32731 in the treatment of psoriasis vulgaris

DETAILED DESCRIPTION:
This is an investigation of the efficacy of LEO 32731 30 mg as compared to placebo after 16 weeks of oral treatment of psoriasis vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Aged between 18 years and 65.
* Males or females of non-childbearing potential.
* Clinical diagnosis of psoriasis vulgaris with or without psoriatic arthritis
* Have moderate to severe psoriasis vulgaris
* Candidates of systemic anti-psoriatic treatment and/or phototherapy

Exclusion Criteria:

* Subjects with therapy resistant psoriasis
* Previously exposed to apremilast
* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris
* Systemic treatment with all other therapies (other than biologics) with a possible effect on psoriasis vulgaris

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) at week 16 | Week 16

SECONDARY OUTCOMES:
Proportion of subjects with Physician's Global Assessment of Disease Severity (PGA) treatment success, defined as clear or almost clear at week 16 | Week 16
Itch evaluated by itch Numerical Rating Scale (NRS) at week 16 | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Philipp, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Dept. of Dermatology, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided